CLINICAL TRIAL: NCT03797365
Title: Randomized Trial to Evaluate the Impact of Cognitive Therapy Added to Normal Perineal Rehabilitation on Pelvic Floor Muscle Contraction for Urinary Incontinent Women.
Brief Title: French Study to Evaluate the Impact of a Cognitive Therapy on Urinary Incontinent Women of All Age's Perineal Settings.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pierre and Marie Curie University (Other)
Collaborators: APHP (Other)
Responsible Party: Principal Investigator, Thubert Thibault, Principal Investigator, Medical Doctor of Gynecology, Pierre and Marie Curie University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cpp17-065a/2016-A01651-50
Record Dates: First submitted 2019-01-02; First posted 2019-01-09 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Urinary Incontinence, Stress; Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: This study is a controlled randomized single blind multicentric study on a sample of 40 women stress or mixed urinary incontinent. Participants will be randomized in two groups with a 1/1 ratio with data processing software at the first visit at the therapist practicing the perineal rehabilitation. The first group will receive "Classical" perineal rehabilitation for duration of height weeks. The second group will receive perineal rehabilitation associated to a double task cognitive therapy for duration of height weeks. Participants will be evaluated during the consultation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical rehabilitation (Active Comparator): Twenty women will benefit from two-phases perineal rehabilitation: first phase pelvic floor muscles (PFM)'s analytic rehabilitation, then a functional rehabilitation.
  Interventions: Other: Classical rehabilitation
- Classical and cognitive associated rehabilitation (Experimental): Twenty women will receive, added to the classic perineal rehabilitation, the cognitive rehabilitation and will have to execute twice a day the rehabilitation protocol.
  Interventions: Behavioral: Cognitive associated rehabilitation

INTERVENTIONS:
Other: Classical rehabilitation — Participants will benefit from two-phases perineal rehabilitation:
  First phase will include the PFM's awareness and voluntary contraction learning with manual, biofeedback technics and functional electro stimulation. These exercises will call out the manual rehabilitation technics, biofeedback and electro stimulation. Each classical rehabilitation session will take 30 minutes with 20 minutes of active working, twice per week. About the self-training, there will be no consensus for optimal homemade exercises.
  For the second phase, a behavior analyze will be summarized in order to update the favoring and inappropriate situations. The strategy put in place will be organized in unlearning of deleterious perineal habits and learning new behavior program. The main goal will be the perineal locking set up, which must be systematic before and during efforts. During this phase, the physiotherapist will twice weekly perform evaluations (similar to those in the first phase)
  Arms: Classical rehabilitation
Behavioral: Cognitive associated rehabilitation — The cognitive associated rehabilitation group randomized participants will have to execute twice a day the rehabilitation protocol. Each cognitive rehabilitation session will take three minutes. Participants will have to synergistically execute attentional tests (N-Back Test) and execute a perineal contraction during the contraction instructions. (10 randomized auditory stimuli in three minutes). The attentional tests' difficulty will be gradually increased each 15 days. N-Back Test modalities are the followings: the participant will visualize a series of random numbers. First difficulty step will be to click the dedicated button when the volunteer will see the indicated letter. The second difficulty step will be to click the dedicated button when she will see two consecutives times the same letter. The third difficulty step will be to click the dedicated button when she will see two times the same letter separated by one different letter, and so on…
  Arms: Classical and cognitive associated rehabilitation

SUMMARY:
This trial is a pathophysiological study evaluating the impact of a cognitive therapy on the perineal neuromuscular mechanisms in women patients with urinary incontinence.

Some research works have been realized on the impact of a cognitive load test (CLT) on the neuromuscular continence urinary mechanisms. It had been demonstrated that a CLT induced an increase in the latency of voluntary perineal contraction. It had also been demonstrated that a CLT had an influence on the involuntary perineal contraction pre-activation. Most recently, the impact of a cognitive therapy on the perineal neuromuscular mechanisms on healthy participants had been evaluated. It demonstrated that a cognitive therapy inhibited the impact of the CLT on the perineal neuromuscular mechanisms.

The present project is about the evaluation of the interest of a cognitive therapy on the neuromuscular mechanisms in case of attentional test in a urinary incontinent women population. It could conduce to new therapeutic leads for the management of urinary incontinence.

DETAILED DESCRIPTION:
Objectives and results expected

Cognition seems to have an effect on the physiological mechanisms of urinary continence. Urinary continence is, among others, the effect of a good coordination between detrusor's contraction and pelvic floor muscles' contraction. A cognitive disturbance involves coordination's disturbance. It has already been demonstrated that a double task rehabilitation (between cognition and perineal muscles) could annihilate the effects induced by a cognitive disturbance on the physiological neuromuscular mechanisms of the urinary incontinence. The objective of this study is to evaluate the benefit of a double task cognitive rehabilitation for the patients with urinary incontinence (UI).

Current knowledge situation

Pelvic floor muscles have a major incidence for the physiological urinary continence. Even if the external anal sphincter (EAS)'s muscles are not directly involved in urinary incontinence, many studies have shown they had a synergistic contraction with levator ani muscles during the voluntary and involuntary perineal contraction . Because they are easily reachable for an electromyographic (EMG) recording, many authors have registered these muscles in order to investigate the physiologic urinary continence. Amarenco et al. had shown that pelvic floor muscles' intensity of contraction in response to a cough fit was proportional to the cough intensity in an healthy volunteers population. This correlation was beyond bladder's filling. For the patients with UI, Deffieux et al. shown a loss of correlation between cough intensity and perineal contraction. Deffieux et al. also analyzed the temporal sequence of muscle activation for the EAS during a cough fit. A perineal pre contraction in an healthy volunteers population was observed. EAS's muscles EMG activation began 210 ms (median) before external intercostal (EIC) muscles. This EAS's muscles anticipation of contraction was not found in the group of patients with UI. The observation that fewer patients were activating their AES's muscles, more the modulation of EAS's muscles contraction was distorted when coughing was made. Thubert et al. observed that the perineal contraction's latency was multiplied by 4 in case of cognitive load test (CLT) in an healthy volunteers population. CLT leads to an EAS's muscles pre activation in case of coughing effort, was also observed. A lowing of 29% of AES's muscles pre activation has been demonstrated. These results suggest that cognition is involved in urinary continence's physiological mechanisms. So it seamed to be interesting to study the impact of a double task rehabilitation (cognitive and muscular) on the urinary continence's neuromuscular mechanisms in case of diversion of attention. It was a randomized trial including two groups of healthy volunteers: one group had double task rehabilitation during 15 days, the other had no rehabilitation. After 15 days rehabilitation, in the rehabilitation's group, the attention deficit's correction restored the resistive abilities of UI in case of attention hijacking.

According to the last AFU's (Association Française d'Urologie - Urology French Association) and CNGOF's (Collège national des gynécologues et obstétriciens français - French Gynecologists and Obstetricians National College) recommendations, the first intention treatment of urinary incontinence is pelvi-perineal rehabilitation. Pelvi-perineal rehabilitation conducted by a therapist is multimodal with different facets: a cognitive part (education, pelvic floor realization), a behavioral part of bladder training (modification of micturition habits), a muscle building part (voluntary contractions against resistance with and without biofeedback and electrosimulation), and also a postural work part (balance and pelvis position). Perineal rehabilitation technics' heterogeneity and the lack of description of these technics let the professionals adapt their rehabilitation's protocols. The objective of this study is to compare the results of two rehabilitation's technics in urinary incontinent patients.

Methodology, study population, previous studies and feasibility

Study population: The population is made of voluntary incontinent women. Inclusion criteria are the followings: Major women with stress urinary incontinence or mixed urinary incontinence or urge urinary incontinence, in need to benefit from perineal rehabilitation or cognitive-behavioral rehabilitation, women able to read, understand, accept and sign the consent. Exclusion criteria are the following: pregnant women, refusal to participate, dementia and cognitive troubles (Mini Mental State score: MMS <30). Participants will be subjects to a medical statement (antecedents, age, weight, size, UDI6 (Urogenital Distress Inventory) questioner, Contilife and Wexner scores). The absence of a mental deficit will be verifies by Mini Mental Status questioner (MMS).

Ethical considerations: A "CPP" (comité de protection des personnes - persons' protection comity) have been requested and obtained for this study (N° cpp17-065a/2016-A01651-50). An information letter will be delivered to the volunteers, who will be included only after the acceptation and signature of the written consent.

Volunteers' randomization: Participants will be randomized in two groups (1/1) with data processing software at the first visit at the therapist practicing the perineal rehabilitation. The first group will receive "Classical" perineal rehabilitation for duration of height weeks. The second group will receive perineal rehabilitation associated with a double task cognitive therapy for a duration of height weeks. Participants will be evaluated during the consultation.

Initial evaluation of volunteers: initial evaluation will consist of an interrogation able to check the participants' antecedents and characteristics, urinary incontinence symptoms (quality life score (Contilife) and severity score (International Consultation on Incontinence Questionnaire Short Form: ICIQ-SF), Urinary Handicap Measurement (MHU - Mesure du Handicap Urinaire) and also clinical examination (Pelvic Organ Prolaps Quantification: POP-Q, Ulmsten Test, levator Testing among Oxford, ureteral mobility). In a second time, the EMG analysis will be realized. It consists in the analysis of the CLT impact on the voluntary and unvoluntary perineal contraction. The CLT used is Paced Auditory Serial addition Test (PASAT). Test arrangements are the followings: The volunteer will listen to an audiotape on witch is recorded a 61 random numbers set inconstant from 1 to 9 (for example "1, 9, 4, 5…"). The volunteer patient will have to add each pair of number in order to add the number with the previous and speak verbally the response. To test the willingly perineal contraction, the volunteer will be in a sitting position with her arms on the armrests. The practitioner will position the two electrodes with self-adhesive surface from either side of the volunteer's anus regarding to the EAS muscle. These electrodes are usually used in a setting of classical evaluation with biofeedback or electro simulation. An order will be given to the volunteer in order to contract perineal muscles when she feels a stimulus on the left wrist (an electric reflex hammer regarding to the median nerve on the inside of the left wrist). The volunteer women will have to repeat the experience in two conditions: with and without the CLT. Different settings measurement will be realized: time limit for the perineal contraction reaction (RT), that is latency between stimulus and begins of AES's EMG activity increase. The other settings will be the RT max (latency between stimulus and maximum AES's EMG activity), maximum AES's EMG activity and air under the curve for the AES's EMG activity. Volunteer's perineal contraction (following coughing instruction) will also be evaluated with and without CLT. The coughing instruction will be ordered by an impulse (Reflex hammer) on the inside of the left wrist. Two more self-adhesive detection electrodes will be glued regarding the external intercostal muscles (7th right space). Principal data analyzed will be: latency between stimulus and perineal muscles (RT1) and latency between intercostal muscles and perineal muscles (RT3). The data set will be collected using a Biopac ®, Acknowledge ®.

Classical perineal rehabilitation protocol

Participants will benefit from two-phases perineal rehabilitation: first phase pelvic floor muscles (PFM)'s analytic rehabilitation, then a functional rehabilitation.

First phase will include the PFM's awareness and voluntary contraction learning with manual, biofeedback technics and functional electro stimulation (FES). Then, therapist will propose PFM's reinforcement under the PERFECT method (Pressure, Endurance, rapid Contraction, time measurement between each contraction sequence). These exercises will call out the manual rehabilitation technics (voluntary contraction learning, pelvic anatomy), biofeedback and electro stimulation. Electro stimulation and biofeedback will necessit the use of an electrode that serves to the electromyographic measurement with and without cognitive load test. Each classical rehabilitation session will take 30 minutes with 20 minutes of active working, twice per week. About the self-training, there will be no consensus for optimal homemade exercises, neither on the number, nor on the duration. The different authors describe very different types of protocols. The self-training program will be set up as soon as the participant will be able to realize, under therapist's manual control, a voluntary analytic contraction without synergy or command reversion. Exercises' number and characteristic will be given according to the PERFECT Scheme.

For the second phase, the participant will hold a micturition calendar. With the noticed elements, a behavior analyze will be summarized in order to update the favoring situations and inappropriate situations. The objective will be the learning of perineal locking and reinstatement of anticipative postural activity for stress urinary incontinence. The strategy put in place will be organized in unlearning of deleterious perineal habits and learning new behavior program. The functional training program will be made of activation of PFM's voluntary contractions during different stains of every day life; the main goal being the perineal locking set up (PFM's voluntary contraction associated with a good abdominal and perineal synergy), this locking must be systematic before and during efforts like carrying loads, trimming, coughing. During the second phase, the physiotherapist will twice weekly perform evaluations. These evaluations are similar to those in the first phase.

Cognitive associated rehabilitation protocol: Added to the classic perineal muscular rehabilitation, the cognitive associated rehabilitation group randomized participants will have to execute twice a day the rehabilitation protocol. Each cognitive rehabilitation session will take three minutes. Participants will have to synergistically execute attentional tests (N-Back Test) and execute a perineal contraction during the contraction instructions. (10 randomized auditory stimuli in three minutes). The attentional tests' difficulty will be gradually increased each 15 days. N-Back Test modalities are the followings: the participant will visualize a series of random numbers. First difficulty step will be to click the dedicated button when the volunteer will see the indicated letter. The second difficulty step will be to click the dedicated button when she will see two consecutives times the same letter. The third difficulty step will be to click the dedicated button when she will see two times the same letter separated by one different letter, and so on… The data will be saved on the digital application.

Methodology: Participants will consult twice per week their therapist. An intermediary clinical and EMG recording will be done in the fourth week to evaluate the evolution of symptoms and EMG's criteria, with the same arrangements as those of the first evaluation.

Participants' final evaluation: During the last visit in the eighth week, participants will be evaluated with same arrangements as those of the first evaluation.

Judgment criteria: About the involuntary perineal contraction study, the principal judgment criteria will be the latency between intercostal muscles contraction and perineal muscles contraction (RT3). Secondary judgment criteria will be: latency between stimulus and perineal muscles contraction (RT1) for the voluntary perineal contraction study, MHU score obtained (Mesure du Handicap Urinaire - urinary handicap score), ICIQ (International Consultation on Incontinence Questionnaire), Contilife.

Statistic analysis:

Descriptive data will be expressed in the form of median and interquartile gap. The Wilcoxon Test will be used to compare quantitative values before and after rehabilitation, and Student Test to compare quantitative values between "classical perineal rehabilitation" group and "perineal rehabilitation + cognitive therapy" group. According to the literature, middle RT3 is -60ms, expected difference after rehabilitation is 16,66ms and known standard deviation is 18,7ms. For an alpha risk 5% and power 80%, it is necessary to include 20 participants by group, whether total of 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* Major women with stress urinary incontinence or mixed urinary incontinence or urge urinary incontinence, in need to benefit from perineal rehabilitation or cognitive-behavioral rehabilitation
* Women able to read, understand, accept and sign the consent.

Exclusion Criteria:

* Pregnant women,
* Refusal to participate
* Dementia and cognitive troubles (MMS<30).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-10 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
RT3 - EMG Latency between intercostal muscles contraction and perineal muscles contraction | Final evaluation at the eighth week follow up
  EMG Latency between intercostal muscles contraction and perineal muscles contraction
RT3 - EMG Latency between intercostal muscles contraction and perineal muscles | Intermediary evaluation at the fourth week follow up
  EMG Latency between intercostal muscles contraction and perineal muscles contraction

SECONDARY OUTCOMES:
RT1 - EMG Latency between stimulus and perineal muscles contraction | Intermediary evaluation at the fourth week follow up, and final evaluation at the eighth week follow up
  EMG Latency between stimulus and perineal muscles contraction
Urinary Handicap Measurement (Mesure du Handicap Urinaire - MHU) | Intermediary evaluation at the fourth week follow up, and final evaluation at the eighth week follow up
  Urinary Handicap Measurement is a quantitative measurement of different urinary symptoms, with 7 different questions, each response is associated to a value from 0 to 4, and with a final score from 0 (lowest score, no symptoms of urinary incontinence) to 28 (Higher score, maximum urinary incontinence symptoms).
International Consultation on Incontinence Questionnaire (ICIQ-SF) | Intermediary evaluation at the fourth week follow up, and final evaluation at the eighth week follow up
  The ICIQ SF is a subjective measurement of severity of urinary loss and quality of life for those with urinary incontinence. It has 4 main items (of 6 total) ask for rating of symptoms in the past 4 weeks. The actual score takes sum score of items 3+4+5 (items 1 and 2 are demographic). The final item (6) is self diagnostic item that is unscored.
  Final score is from 0 (lowest score, no symptoms of urinary incontinence), to 21 (Higher score, maximum urinary incontinence symptoms).
Questionnaire for assessment of quality of life related to women urinary incontinence (Contilife) | Intermediary evaluation at the fourth week follow up, and final evaluation at the eighth week follow up
  Auto survey of 28 questions for the quality of life related to the women with urinary incontinence. There are 6 main subjects related to quality of life, and each question has a score from 0 or 1 to 5. The final score is Final score is from 23 (lowest score, no impact of urinary incontinence on quality of life), to 140 (Higher score, maximum impact of urinary incontinence on quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Thibault THUBERT, MD, Principal Investigator — CHU Hotel Dieu Nantes; Pierre-André MAL, resident, Study Chair — CHU Hopital Tenon APHP

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sapsford RR, Hodges PW. Contraction of the pelvic floor muscles during abdominal maneuvers. Arch Phys Med Rehabil. 2001 Aug;82(8):1081-8. doi: 10.1053/apmr.2001.24297. PMID 11494188
- [Background] Amarenco G, Ismael SS, Lagauche D, Raibaut P, Rene-Corail P, Wolff N, Thoumie P, Haab F. Cough anal reflex: strict relationship between intravesical pressure and pelvic floor muscle electromyographic activity during cough. Urodynamic and electrophysiological study. J Urol. 2005 Jan;173(1):149-52. doi: 10.1097/01.ju.0000147305.00443.df. PMID 15592060
- [Background] Deffieux X, Hubeaux K, Porcher R, Ismael SS, Raibaut P, Amarenco G. External intercostal muscles and external anal sphincter electromyographic activity during coughing. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Apr;19(4):521-4. doi: 10.1007/s00192-007-0473-y. Epub 2007 Oct 13. PMID 17934686
- [Background] Fritel X, Fauconnier A, Bader G, Cosson M, Debodinance P, Deffieux X, Denys P, Dompeyre P, Faltin D, Fatton B, Haab F, Hermieux JF, Kerdraon J, Mares P, Mellier G, Michel-Laaengh N, Nadeau C, Robain G, de Tayrac R, Jacquetin B; French College of Gynaecologists and Obstetricians. Diagnosis and management of adult female stress urinary incontinence: guidelines for clinical practice from the French College of Gynaecologists and Obstetricians. Eur J Obstet Gynecol Reprod Biol. 2010 Jul;151(1):14-9. doi: 10.1016/j.ejogrb.2010.02.041. Epub 2010 Mar 16. PMID 20236751
- [Background] Hermieu JF, Denys P, Fritel X. [Critical review of guidelines for female urinary incontinence diagnosis and treatment]. Prog Urol. 2012 Oct;22(11):636-43. doi: 10.1016/j.purol.2012.08.004. Epub 2012 Sep 10. French. PMID 22999088
- [Background] Klovning A, Avery K, Sandvik H, Hunskaar S. Comparison of two questionnaires for assessing the severity of urinary incontinence: The ICIQ-UI SF versus the incontinence severity index. Neurourol Urodyn. 2009;28(5):411-5. doi: 10.1002/nau.20674. PMID 19214996
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Background] Horton AM Jr, Alana S. Validation of the Mini-Mental State Examination. Int J Neurosci. 1990 Aug;53(2-4):209-12. doi: 10.3109/00207459008986604. PMID 2265941
- [Result] Thubert T, Villot A, Billecocq S, Auclair L, Amarenco G, Deffieux X. Influence of a distraction task on the involuntary reflex contraction of the pelvic floor muscles following cough. Neurourol Urodyn. 2017 Jan;36(1):160-165. doi: 10.1002/nau.22903. Epub 2015 Oct 9. PMID 26451967
- [Result] Thubert T, Deffieux X, Jousse M, Guinet-Lacoste A, Ismael SS, Amarenco G. Influence of a distraction task on pelvic floor muscle contraction. Neurourol Urodyn. 2015 Feb;34(2):139-43. doi: 10.1002/nau.22524. Epub 2014 Feb 12. PMID 24519688
- [Result] Villot A, Deffieux X, Billecocq S, Auclair L, Amarenco G, Thubert T. Influence of cognitive rehabilitation on pelvic floor muscle contraction: A randomized controlled trial. Neurourol Urodyn. 2017 Aug;36(6):1636-1644. doi: 10.1002/nau.23169. Epub 2016 Oct 29. PMID 27794195
- [Result] Deffieux X, Hubeaux K, Porcher R, Ismael SS, Raibaut P, Amarenco G. Pelvic floor muscle activity during coughing: altered pattern in women with stress urinary incontinence. Urology. 2007 Sep;70(3):443-7; discussion 447-8. doi: 10.1016/j.urology.2007.03.084. PMID 17905093
- [Result] Deffieux X, Hubeaux K, Porcher R, Ismael SS, Raibaut P, Amarenco G. Abnormal pelvic response to cough in women with stress urinary incontinence. Neurourol Urodyn. 2008;27(4):291-6. doi: 10.1002/nau.20506. PMID 17803192